CLINICAL TRIAL: NCT03616353
Title: IMpact of Perineural Hydrodissection Over Alternative Therapies in Patients With Carpal Tunnel Syndrome (IMPACTS): A Single-Centre, Randomized Trial Comparing Perineural Hydrodissection of the Median Nerve Versus Steroid Injection in Patients With Carpal Tunnel Syndrome
Brief Title: IMpact of Perineural Hydrodissection Over Alternative Therapies in Patients With Carpal Tunnel Syndrome
Acronym: IMPACTS
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leslie Witton (Other)
Responsible Party: Sponsor-Investigator, Leslie Witton, Neurology Resident, Hamilton Health Sciences Corporation
Organization: Hamilton Health Sciences Corporation (Other)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2017-07-31; First posted 2018-08-06 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Adrenal Cortex Hormones; Steroids

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Care provider is performing a specific type of injection and therefore cannot be blinded. Those investigators responsible for collecting, managing, and analyzing data will be blinded to treatment randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Corticosteroid Injection (Experimental): Patients in this group will undergo an injection of corticosteroid into the carpal tunnel as per current treatment practices.
  Interventions: Procedure: Corticosteroid Injection
- Group 2: Perineural Hydrodissection (Experimental): Patients in this group will undergo a perineural hydrodissection plus an injection of corticosteroid into the carpal tunnel, as a novel technique.
  Interventions: Procedure: Perineural Hydrodissection

INTERVENTIONS:
Procedure: Perineural Hydrodissection — The subcutaneous tissues of the ulnar aspect of the wrist at the level of the carpal tunnel will be infiltrated with 2 ml of lidocaine 1% for local anesthetic. Using ultrasound guidance and aseptic technique, the needle will then be angled deep to the median nerve within the carpal tunnel, and 5 ml of a 50%/50% mixture of lidocaine 1% and sensorcaine 0.5% will be injected under pressure. While continuing to use ultrasound guidance and aseptic technique, the needle will then be angled superficial to the median nerve within the carpal tunnel, and 5 ml of a 50%/50% mixture of lidocaine 1% and sensorcaine 0.5% will be injected under pressure. The needle will be returned to its original angle deep to the median nerve, and the syringe will be changed to inject 40 mg Depo-Medrol in 1ml of saline.
  Other Names: PNH
  Arms: Group 2: Perineural Hydrodissection
Procedure: Corticosteroid Injection — The subcutaneous soft tissues of the ulnar aspect of the wrist at the level of the carpal tunnel will be infiltrated with 2 ml of lidocaine 1% for local anesthetic. Using ultrasound guidance and aseptic technique, the needle will then be angled deep to the median nerve within the carpal tunnel, and 40 mg Depo-Medrol in 1ml of saline will be injected into the area deep to the median nerve.
  Other Names: Steroid
  Arms: Group 1: Corticosteroid Injection

SUMMARY:
This is a multidisciplinary, single-blinded, three-arm randomized controlled trial, comparing perineural hydrodissection and steroid injection for the treatment of CTS. Patients are screened based on pre-established eligibility criteria and randomized to one of the three study groups. Patients are followed at 6-week, 3-month, 6-month, and 12-month time points to assess the primary and secondary outcomes of the study, which include both patient-reported outcome measures and objective clinical assessments.

DETAILED DESCRIPTION:
This study aims to examine the effect of perineural hydrodissection (PNH), a novel treatment for CTS. PNH is a minimally invasive, ultrasound-guided, percutaneous technique in which the median nerve is released by injecting fluid (local anesthetic and corticosteroid) circumferentially, using larger fluid volumes and higher pressure to target areas of adhesion between the median nerve and its surrounding structures. In chronic CTS, a rind of perineural fibrosis develops, tethering the median nerve to the overlying flexor retinaculum and to the adjacent flexor tendons. Theoretically, the removal of tethering to adjacent structures, via perineural hydrodissection, should allow circumferential bathing of the median nerve with the local anesthetic and corticosteroid, thus reducing inflammation and prolonging symptom relief.

The primary outcome is pain as measured by the Boston Carpal Tunnel Questionnaire (BCTQ). Secondary outcomes include health-related quality of life measures using the Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire and the Visual Analog Scale (VAS) for pain.

The selected questionnaires have been shown to correlate well with domains of the International Classification of Functioning, Disability, and Health (ICF) (3). Other secondary measures include the ultrasound appearance (cross-sectional index) of the median nerve, and electromyography (EMG) measurements (including sensory and motor conduction velocities, and amplitudes), before and after the injection.

The study hypothesis is that PNH will show greater benefits in terms of pain, function, and patient quality of life when compared to corticosteroid injection in patients with CTS. The null hypothesis is that there is no difference. The study is powered to address the primary outcome and will also be powered to identify minimally important differences in functional, sonographic, and electromyographic outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men or women aged 18 years or greater.
2. Clinical and electromyographic diagnosis of Carpal Tunnel Syndrome.
3. Persistent symptoms from Carpal Tunnel Syndrome after at least three months of appropriate splinting.
4. Ability to consent for study.

Exclusion Criteria:

1. Acute symptom onset (less than 3 months).
2. Bifid median nerve
3. Anticoagulation with International Normalized Ratio (INR) > 1.4, or platelets <150.
4. Anomalous muscles (eg. inverted palmaris longus).
5. Patients requiring anti-platelet medication for the treatment of heart attack, stroke, or other medical condition.
6. Previous surgery for Carpal Tunnel Syndrome.
7. Previous local injections, including steroids within the past 6 months.
8. Allergy to any of the injection agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Boston Carpal Tunnel Questionnaire (BCTQ) | Baseline, 6 weeks, 3 months, 6 months, 1 year
  The BCTQ is a five-point rating scale with 19 items. The overall score is the average score across all items. The score will be recorded for each visit and change in score will be plotted over time.

SECONDARY OUTCOMES:
Change in Ultrasonographic Measurement | Baseline, 6 weeks, 6 months, 1 year
  Cross-sectional index (CSI) of the median nerve as measured by ultrasound. The CSI will be recorded for each visit and change will be plotted over time.
Change in Electromyographic Measurement- Amplitude | Baseline, 6 months, 1 year
  Amplitudes will be recorded for each visit and change in these values will be plotted over time.
Change in Electromyographic Measurement- Motor Conduction Velocity | Baseline, 6 months, 1 year
  Motor conduction velocities will be recordedfor each visit and change in these values will be plotted over time.
Change in Electromyographic Measurement- Sensory Conduction Velocity | Baseline, 6 months, 1 year
  Sensory conduction velocities will be recordedfor each visit and change in these values will be plotted over time.
Change in Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire | Baseline, 6 weeks, 3 months, 6 months, 1 year
  The DASH is a 30-item measure using five-point Likert scales assessing aspects of physical functioning and symptoms, intended specifically to measure disability. Its overall score is between 0 and 100. The score will be recorded for each visit and change in score will be plotted over time.
Change in Visual Analog Scale (VAS) for Pain | Baseline, 6 weeks, 3 months, 6 months, 1 year
  The VAS is a commonly used, subjective scale in which the patient rates their pain on a scale ranging from 0 to 10 (0, no pain; 10, maximum pain possible). The score will be recorded for each visit and change will be plotted over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Hamilton Health Sciences, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No